CLINICAL TRIAL: NCT05681416
Title: Prostate Cancer Prevention Clinic for Men With Risk of Familial Prostate Cancer
Acronym: ProFam-Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Principal Investigator, Jale Lakes, senior doctor at the department of urology, Heinrich-Heine University, Duesseldorf
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Studien-Nr.: 2022-2051
Record Dates: First submitted 2022-11-29; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer; Familial Prostate Cancer
Keywords: BRCA Mutation; Familial Prostate Cancer; Genetic Predisposition; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Prostate cancer, familial; Genetic Predisposition to Disease | interventions — Exome; Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Men with family history or already known BRCA1 or BRCA2 mutation and their family members will be offered a combined clinical, imaging and genetic profiling to tailor their risk to develop PCA. In addition, men with prostate cancer and positive family history will be offered genetic testing and mutational profiling of tumor tissue in order to exclude or detect hereditary cancer syndromes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy men with familial risk (Other): ≥ 2 first-degree relatives with PCA diagnosed at any age oder ≥ 1 first-degree relative with PCA diagnosed at the age <60
  Interventions: Diagnostic Test: Panel sequencing, whole exome sequencing, whole genome sequencing
- healthy men with genetic risk (Other): BRCA1/2 Germline mutation
  Interventions: Diagnostic Test: Panel sequencing, whole exome sequencing, whole genome sequencing
- Men with PCA and genetic oder familial risk (Other): familial risk = ≥ 2 first-degree relatives with PCA diagnosed at any age oder ≥ 1 first-degree relative with PCA diagnosed at the age <60 genetic risk= BRCA1/2 Germline mutation
  Interventions: Diagnostic Test: Panel sequencing, whole exome sequencing, whole genome sequencing

INTERVENTIONS:
Diagnostic Test: Panel sequencing, whole exome sequencing, whole genome sequencing — Besides the mutation positive men (group 2), all will receive multigene panel analysis in a patient care setting and if negative, whole exome sequencing (WES), whole genome sequencing and transcriptome analyses. In PCA-affected men (group 3), additional mutational analysis will be performed on formalin-fixed paraffin embedded (FFPE) - and fresh frozen (FF) tumor tissue from biobanked radical prostatectomy specimens using FFPE panel analysis (like TruSightOncology 500) or WES if FF samples are available.
  Other Names: mpMRI; psychometric tests; PSA Testing

SUMMARY:
Secondary prevention of prostate cancer (PCa) is not standardized and high-risk groups at the time of diagnosis are not well defined. Hereditary susceptibility which is reported in about 10% of men is one important risk factor for PCa development but the absolute risk and clinical importance is fairly unknown. The population risk for developing PCa is estimated to be 11%. If men carry a mutation in BRCA2 or HOXB13, the lifetime risk is 2 to 10-fold increased. "ProFam-Risk" is a prospective cohort analysis not only to validate the known genetic risk scores but also to establish recommendations for follow of high risk populations based on a combination of clinical parameters, imaging (magnetic resonance imaging of the prostate), and genetic profile. Aim of this individualized recommendation is on the one hand to early detect PCa before developing of advanced disease and on the other hand to counsel men at low risk in order to prevent overdiagnosis and overtreatment. Overall, "ProFam-Risk" aims to create a best possible counseling and clinical care for men with familial risk to develop PCa. In this pilot study, about 100 men per year will be included for a total period of 3 years. In addition to the registration of clinical, imaging, and genetic information, liquids and tissue (if available) will be sampled for analysis in the above mentioned research questions.

DETAILED DESCRIPTION:
Prostate cancer (PCA) is common in men. If men carry a mutation in BRCA2 or HOXB13, the lifetime risk is 2 to 10-fold increased. Germline testing is used for individualized risk prediction. In the context of the precision medicine era, different multigene panels are used for hereditary cancer syndromes, including hereditary breast and ovarian cancer (HBOC), Lynch syndrome and hereditary prostate cancer . In addition, targeted therapy with e.g. PARP inhibitors and immunotherapeutic drugs is based on the presence of mutations in DNA repair genes such as BRCA1 and BRCA2, ATM or mismatch repair genes . Furthermore, polygenic risk scores (PRS) are associated with the risk to develop prostate cancer in European and multi-ethnic ancestries with HRs of 1.6 to 5 . Trans-ancestry genome-wide association studies have revealed 269 risk variants from tissue related to prostate cancer including known tumor-related genes like TP53 and CHEK2 .

To more precisely tailor screening for prostate cancer, risk groups with a higher prevalence of clinically significant PCA (csPCA) need to be defined.

Current NCCN guidelines recommend e. g. genetic testing for men with a positive family history of PCA. The prevalence of germline variants in these men diagnosed with PCA at age 60 was 17.2% of which about 30% were BRCA1 or BRCA2 mutations and 4.5% were HOXB13. The absolute risk to develop PCA up to the age of 80 years in BRCA2 carriers is supposed to be 27% - 60%.

Limited data are available concerning the mutational landscape of PCA and somatic oncogenic drivers. To date, studies predominantly focused on known tumor genes with potential clinical actionability and their underlying pathways to guide clinical management in advanced tumor diseases. Systematic mutational profiling in different stages of tumor disease and correlation with germline findings are urgently needed for an in depth understanding of the prostate cancer pathogenesis and identifying promising drug candidates as well as early detection of driver mutations for lethal cancers.

First attempts to combine clinical and genetic data are currently tested in the PROFILE and BARCODE 1 studies. Men with a positive family history of PCA at age 40-69 years were recommended to undergo prostate biopsy regardless of prostate specific antigen (PSA) levels and 25% of those had PCA. The succeeding BARCODE 1 trial is currently recruiting men at ages 55-69 years who are offered genotyping by 130 germline PCA risk single nucleotide polymorphisms (SNPs) from saliva. After calculating a polygenic risk score (PRS), participants above the 90% percentile are offered screening by magnetic resonance imaging (MRI) followed by prostate biopsy. Prostate cancer detection was about 40% of all men screened within the pilot study.

Multiparametric MRI (mpMRI) was developed and explored in prospective and randomized trials also within the group in Düsseldorf to personalize the indication for a prostate biopsy. In collaboration with international partners, mpMRI was shown to improve the accuracy of PCA detection. In addition, the Düsseldorf branch of the hereditary breast and ovarian cancer (HBOC) consortium was part of an international analysis of non-HBOC cancer risks in BRCA1 and BRCA2 mutation carriers. By this analysis, more than 50 men with BRCA2 mutation were identified in the Düsseldorf cohort alone.

Within the National Cancer Prevention Graduate School, the German Cancer Aid (DKH) lately funded the newly established Prostate Cancer Prevention Clinic for men with familial risk at Düsseldorf University. This is a unique and first of its kind outpatient clinic which will include about 100 men at risk for PCA per year and offer specialized diagnostics as a combination of multiparametric MRI, psychometric tests, and genetic analysis to establish an individualized risk score with consecutive risk-adapted monitoring. Men with family history or already known BRCA1 or BRCA2 mutation and their family members will be offered a combined clinical, imaging and genetic profiling to tailor their risk to develop PCA. In addition, men with prostate cancer and positive family history will be offered genetic testing and mutational profiling of tumor tissue in order to exclude or detect hereditary cancer syndromes.

The overarching goal of this project is to identify novel cancer signaling pathways based on the identification of previously unreported genes causative for PCA and to extract preventive and therapeutic approaches for PCA . The groundwork is the establishment of a prospective cohort of unaffected men with a higher risk for PCA due to PCA affected family members ("index patients") (group 1) and/or a mutation in the BRCA1/2 genes (group 2) and PCA-affected men (group 3) . Besides the mutation positive men (group 2) , all will receive multigene panel analysis in a patient care setting and if negative, whole exome sequencing (WES), whole genome sequencing and transcriptome analyses. In PCA-affected men (group 3), additional mutational analysis will be performed on formalin-fixed paraffin embedded (FFPE) - and fresh frozen (FF) tumor tissue from biobanked radical prostatectomy specimens using FFPE panel analysis or WES if FF samples are available.

The investigators propose the following aims:

1. Assembly and clinical characterization of a prospective PCA cohort
2. Identification of PCA-related gene alterations in novel genes
3. Genotype-phenotype correlations and prevention of overdiagnosis/overtreatment by risk-adapted individualized follow-up investigations

ELIGIBILITY:
Inclusion criteria:

* Healthy men with familial risk ( ≥ 2 first-degree relatives with PCA diagnosed at any age oder ≥ 1 first-degree relative with PCA diagnosed at the age <60)
* healthy men with genetic risk (BRCA1/2 Germline mutation)
* Men with PCA and genetic oder familial risk (familial risk = ≥ 2 first-degree relatives with PCA diagnosed at any age oder ≥ 1 first-degree relative with PCA diagnosed at the age <60; genetic risk= BRCA1/2 Germline mutation)

Exclusion criteria:

* <18 years
* no consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is only observed in men
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Number and kind of Genetic Alterations and correlation with clinical and pathologic features | 3-4 years
  mutation database for germline mutations and tumor mutations in familial PCA:
  Besides the mutation positive men (group 2), all will receive multigene panel analysis( ATM, BRCA1, BRCA2, EPCAM, HOXB13, MLH1, MSH2, MSH6, PMS2, TP53) and if negative, whole exome sequencing (WES), whole genome sequencing and transcriptome analyses The aim is to systematically and prospektively review genotype-phenotype correlations in the established candidate genes and to systematically correlate the clinical and pathologic features with the identified underlying genetic alterations.
  DNA for WES, WGS and RNA will be prepared by standard procedures, e.g. the FlexiGene DNA Kit (Qiagen) and PAXgene Blood RNA Kit (Qiagen)
Reduction in PCA-specific anxiety | 3-4 years
  Assessment if men after risk assessment and genetic counseling will have a reduction in cancer-specific anxiety -->Follow-ups with 3 measurement points (before, during, after counseling (T0, T1, T2)) The reduction in cancer-specific anxiety and improvement of personal risk perception and of personal control are tested by using a of variance- analytical model with repeated measures (T0, T1, T2) and the group factor "risk group" (high vs. intermediate vs. low)
  Quantitative questionnaire:
  • Prostate Cancer-specific anxiety (MAX-PC, modified scale 'prostate cancer anxiety', Lehmann 2006)

SECONDARY OUTCOMES:
Improvement of PCA-specific personal risk perception | 3-4 years
  Assessment if men after risk assessment and genetic counseling will have an improvement of PCA-specific personal risk perception
  -->Follow-ups with 3 measurement points (before, during, after counseling (T0, T1, T2)) The improvement of personal risk perception are tested by using a of variance- analytical model with repeated measures (T0, T1, T2) and the group factor "risk group" (high vs. intermediate vs. low)
  Quantitative questionnaire:
  • Risk perception of prostate cancer (Shavers 2009)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Albers, Principal Investigator — Department of Urology, University of Dusseldorf, Germany; Dagmar Wieczorek, Principal Investigator — Humangenetics, University of Dusseldorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li S, Silvestri V, Leslie G, Rebbeck TR, Neuhausen SL, Hopper JL, Nielsen HR, Lee A, Yang X, McGuffog L, Parsons MT, Andrulis IL, Arnold N, Belotti M, Borg A, Buecher B, Buys SS, Caputo SM, Chung WK, Colas C, Colonna SV, Cook J, Daly MB, de la Hoya M, de Pauw A, Delhomelle H, Eason J, Engel C, Evans DG, Faust U, Fehm TN, Fostira F, Fountzilas G, Frone M, Garcia-Barberan V, Garre P, Gauthier-Villars M, Gehrig A, Glendon G, Goldgar DE, Golmard L, Greene MH, Hahnen E, Hamann U, Hanson H, Hassan T, Hentschel J, Horvath J, Izatt L, Janavicius R, Jiao Y, John EM, Karlan BY, Kim SW, Konstantopoulou I, Kwong A, Lauge A, Lee JW, Lesueur F, Mebirouk N, Meindl A, Mouret-Fourme E, Musgrave H, Ngeow Yuen Yie J, Niederacher D, Park SK, Pedersen IS, Ramser J, Ramus SJ, Rantala J, Rashid MU, Reichl F, Ritter J, Rump A, Santamarina M, Saule C, Schmidt G, Schmutzler RK, Senter L, Shariff S, Singer CF, Southey MC, Stoppa-Lyonnet D, Sutter C, Tan Y, Teo SH, Terry MB, Thomassen M, Tischkowitz M, Toland AE, Torres D, Vega A, Wagner SA, Wang-Gohrke S, Wappenschmidt B, Weber BHF, Yannoukakos D, Spurdle AB, Easton DF, Chenevix-Trench G, Ottini L, Antoniou AC. Cancer Risks Associated With BRCA1 and BRCA2 Pathogenic Variants. J Clin Oncol. 2022 May 10;40(14):1529-1541. doi: 10.1200/JCO.21.02112. Epub 2022 Jan 25. PMID 35077220
- [Background] Ewing CM, Ray AM, Lange EM, Zuhlke KA, Robbins CM, Tembe WD, Wiley KE, Isaacs SD, Johng D, Wang Y, Bizon C, Yan G, Gielzak M, Partin AW, Shanmugam V, Izatt T, Sinari S, Craig DW, Zheng SL, Walsh PC, Montie JE, Xu J, Carpten JD, Isaacs WB, Cooney KA. Germline mutations in HOXB13 and prostate-cancer risk. N Engl J Med. 2012 Jan 12;366(2):141-9. doi: 10.1056/NEJMoa1110000. PMID 22236224
- [Background] Russo J, Giri VN. Germline testing and genetic counselling in prostate cancer. Nat Rev Urol. 2022 Jun;19(6):331-343. doi: 10.1038/s41585-022-00580-7. Epub 2022 Apr 21. PMID 35449224
- [Background] Barnes DR, Silvestri V, Leslie G, McGuffog L, Dennis J, Yang X, Adlard J, Agnarsson BA, Ahmed M, Aittomaki K, Andrulis IL, Arason A, Arnold N, Auber B, Azzollini J, Balmana J, Barkardottir RB, Barrowdale D, Barwell J, Belotti M, Benitez J, Berthet P, Boonen SE, Borg A, Bozsik A, Brady AF, Brennan P, Brewer C, Brunet J, Bucalo A, Buys SS, Caldes T, Caligo MA, Campbell I, Cassingham H, Christensen LL, Cini G, Claes KBM; GEMO Study Collaborators; EMBRACE Collaborators; Cook J, Coppa A, Cortesi L, Damante G, Darder E, Davidson R, de la Hoya M, De Leeneer K, de Putter R, Del Valle J, Diez O, Ding YC, Domchek SM, Donaldson A, Eason J, Eeles R, Engel C, Evans DG, Feliubadalo L, Fostira F, Frone M, Frost D, Gallagher D, Gehrig A, Giraud S, Glendon G, Godwin AK, Goldgar DE, Greene MH, Gregory H, Gross E, Hahnen E, Hamann U, Hansen TVO, Hanson H, Hentschel J, Horvath J; KConFab Investigators; HEBON Investigators; Izatt L, Izquierdo A, James PA, Janavicius R, Jensen UB, Johannsson OT, John EM, Kramer G, Kroeldrup L, Kruse TA, Lautrup C, Lazaro C, Lesueur F, Lopez-Fernandez A, Mai PL, Manoukian S, Matrai Z, Matricardi L, Maxwell KN, Mebirouk N, Meindl A, Montagna M, Monteiro AN, Morrison PJ, Muranen TA, Murray A, Nathanson KL, Neuhausen SL, Nevanlinna H, Nguyen-Dumont T, Niederacher D, Olah E, Olopade OI, Palli D, Parsons MT, Pedersen IS, Peissel B, Perez-Segura P, Peterlongo P, Petersen AH, Pinto P, Porteous ME, Pottinger C, Pujana MA, Radice P, Ramser J, Rantala J, Robson M, Rogers MT, Ronlund K, Rump A, Sanchez de Abajo AM, Shah PD, Sharif S, Side LE, Singer CF, Stadler Z, Steele L, Stoppa-Lyonnet D, Sutter C, Tan YY, Teixeira MR, Teule A, Thull DL, Tischkowitz M, Toland AE, Tommasi S, Toss A, Trainer AH, Tripathi V, Valentini V, van Asperen CJ, Venturelli M, Viel A, Vijai J, Walker L, Wang-Gohrke S, Wappenschmidt B, Whaite A, Zanna I, Offit K, Thomassen M, Couch FJ, Schmutzler RK, Simard J, Easton DF, Chenevix-Trench G, Antoniou AC, Ottini L; Consortium of Investigators of Modifiers of BRCA1 and BRCA2. Breast and Prostate Cancer Risks for Male BRCA1 and BRCA2 Pathogenic Variant Carriers Using Polygenic Risk Scores. J Natl Cancer Inst. 2022 Jan 11;114(1):109-122. doi: 10.1093/jnci/djab147. PMID 34320204
- [Background] Conti DV, Darst BF, Moss LC, Saunders EJ, Sheng X, Chou A, Schumacher FR, Olama AAA, Benlloch S, Dadaev T, Brook MN, Sahimi A, Hoffmann TJ, Takahashi A, Matsuda K, Momozawa Y, Fujita M, Muir K, Lophatananon A, Wan P, Le Marchand L, Wilkens LR, Stevens VL, Gapstur SM, Carter BD, Schleutker J, Tammela TLJ, Sipeky C, Auvinen A, Giles GG, Southey MC, MacInnis RJ, Cybulski C, Wokolorczyk D, Lubinski J, Neal DE, Donovan JL, Hamdy FC, Martin RM, Nordestgaard BG, Nielsen SF, Weischer M, Bojesen SE, Roder MA, Iversen P, Batra J, Chambers S, Moya L, Horvath L, Clements JA, Tilley W, Risbridger GP, Gronberg H, Aly M, Szulkin R, Eklund M, Nordstrom T, Pashayan N, Dunning AM, Ghoussaini M, Travis RC, Key TJ, Riboli E, Park JY, Sellers TA, Lin HY, Albanes D, Weinstein SJ, Mucci LA, Giovannucci E, Lindstrom S, Kraft P, Hunter DJ, Penney KL, Turman C, Tangen CM, Goodman PJ, Thompson IM Jr, Hamilton RJ, Fleshner NE, Finelli A, Parent ME, Stanford JL, Ostrander EA, Geybels MS, Koutros S, Freeman LEB, Stampfer M, Wolk A, Hakansson N, Andriole GL, Hoover RN, Machiela MJ, Sorensen KD, Borre M, Blot WJ, Zheng W, Yeboah ED, Mensah JE, Lu YJ, Zhang HW, Feng N, Mao X, Wu Y, Zhao SC, Sun Z, Thibodeau SN, McDonnell SK, Schaid DJ, West CML, Burnet N, Barnett G, Maier C, Schnoeller T, Luedeke M, Kibel AS, Drake BF, Cussenot O, Cancel-Tassin G, Menegaux F, Truong T, Koudou YA, John EM, Grindedal EM, Maehle L, Khaw KT, Ingles SA, Stern MC, Vega A, Gomez-Caamano A, Fachal L, Rosenstein BS, Kerns SL, Ostrer H, Teixeira MR, Paulo P, Brandao A, Watya S, Lubwama A, Bensen JT, Fontham ETH, Mohler J, Taylor JA, Kogevinas M, Llorca J, Castano-Vinyals G, Cannon-Albright L, Teerlink CC, Huff CD, Strom SS, Multigner L, Blanchet P, Brureau L, Kaneva R, Slavov C, Mitev V, Leach RJ, Weaver B, Brenner H, Cuk K, Holleczek B, Saum KU, Klein EA, Hsing AW, Kittles RA, Murphy AB, Logothetis CJ, Kim J, Neuhausen SL, Steele L, Ding YC, Isaacs WB, Nemesure B, Hennis AJM, Carpten J, Pandha H, Michael A, De Ruyck K, De Meerleer G, Ost P, Xu J, Razack A, Lim J, Teo SH, Newcomb LF, Lin DW, Fowke JH, Neslund-Dudas C, Rybicki BA, Gamulin M, Lessel D, Kulis T, Usmani N, Singhal S, Parliament M, Claessens F, Joniau S, Van den Broeck T, Gago-Dominguez M, Castelao JE, Martinez ME, Larkin S, Townsend PA, Aukim-Hastie C, Bush WS, Aldrich MC, Crawford DC, Srivastava S, Cullen JC, Petrovics G, Casey G, Roobol MJ, Jenster G, van Schaik RHN, Hu JJ, Sanderson M, Varma R, McKean-Cowdin R, Torres M, Mancuso N, Berndt SI, Van Den Eeden SK, Easton DF, Chanock SJ, Cook MB, Wiklund F, Nakagawa H, Witte JS, Eeles RA, Kote-Jarai Z, Haiman CA. Trans-ancestry genome-wide association meta-analysis of prostate cancer identifies new susceptibility loci and informs genetic risk prediction. Nat Genet. 2021 Jan;53(1):65-75. doi: 10.1038/s41588-020-00748-0. Epub 2021 Jan 4. PMID 33398198
- [Background] Mohler JL, Antonarakis ES, Armstrong AJ, D'Amico AV, Davis BJ, Dorff T, Eastham JA, Enke CA, Farrington TA, Higano CS, Horwitz EM, Hurwitz M, Ippolito JE, Kane CJ, Kuettel MR, Lang JM, McKenney J, Netto G, Penson DF, Plimack ER, Pow-Sang JM, Pugh TJ, Richey S, Roach M, Rosenfeld S, Schaeffer E, Shabsigh A, Small EJ, Spratt DE, Srinivas S, Tward J, Shead DA, Freedman-Cass DA. Prostate Cancer, Version 2.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 May 1;17(5):479-505. doi: 10.6004/jnccn.2019.0023. PMID 31085757
- [Background] Nyberg T, Frost D, Barrowdale D, Evans DG, Bancroft E, Adlard J, Ahmed M, Barwell J, Brady AF, Brewer C, Cook J, Davidson R, Donaldson A, Eason J, Gregory H, Henderson A, Izatt L, Kennedy MJ, Miller C, Morrison PJ, Murray A, Ong KR, Porteous M, Pottinger C, Rogers MT, Side L, Snape K, Walker L, Tischkowitz M, Eeles R, Easton DF, Antoniou AC. Prostate Cancer Risks for Male BRCA1 and BRCA2 Mutation Carriers: A Prospective Cohort Study. Eur Urol. 2020 Jan;77(1):24-35. doi: 10.1016/j.eururo.2019.08.025. Epub 2019 Sep 6. PMID 31495749
- [Background] Castro E, Mikropoulos C, Bancroft EK, Dadaev T, Goh C, Taylor N, Saunders E, Borley N, Keating D, Page EC, Saya S, Hazell S, Livni N, deSouza N, Neal D, Hamdy FC, Kumar P, Antoniou AC, Kote-Jarai Z; PROFILE Study Steering Committee; Eeles RA. The PROFILE Feasibility Study: Targeted Screening of Men With a Family History of Prostate Cancer. Oncologist. 2016 Jun;21(6):716-22. doi: 10.1634/theoncologist.2015-0336. Epub 2016 May 5. PMID 27151655
- [Background] Benafif S, Ni Raghallaigh H, McGrowder E, Saunders EJ, Brook MN, Saya S, Rageevakumar R, Wakerell S, James D, Chamberlain A, Taylor N, Hogben M, Benton B, D'Mello L, Myhill K, Mikropoulos C, Bowen-Perkins H, Rafi I, Ferris M, Beattie A, Kuganolipava S, Sevenoaks T, Bower J, Kumar P, Hazell S, deSouza NM, Antoniou A, Bancroft E, Kote-Jarai Z, Eeles R. The BARCODE1 Pilot: a feasibility study of using germline single nucleotide polymorphisms to target prostate cancer screening. BJU Int. 2022 Mar;129(3):325-336. doi: 10.1111/bju.15535. Epub 2021 Aug 15. PMID 34214236
- [Background] Giri VN, Knudsen KE, Kelly WK, Cheng HH, Cooney KA, Cookson MS, Dahut W, Weissman S, Soule HR, Petrylak DP, Dicker AP, AlDubayan SH, Toland AE, Pritchard CC, Pettaway CA, Daly MB, Mohler JL, Parsons JK, Carroll PR, Pilarski R, Blanco A, Woodson A, Rahm A, Taplin ME, Polascik TJ, Helfand BT, Hyatt C, Morgans AK, Feng F, Mullane M, Powers J, Concepcion R, Lin DW, Wender R, Mark JR, Costello A, Burnett AL, Sartor O, Isaacs WB, Xu J, Weitzel J, Andriole GL, Beltran H, Briganti A, Byrne L, Calvaresi A, Chandrasekar T, Chen DYT, Den RB, Dobi A, Crawford ED, Eastham J, Eggener S, Freedman ML, Garnick M, Gomella PT, Handley N, Hurwitz MD, Izes J, Karnes RJ, Lallas C, Languino L, Loeb S, Lopez AM, Loughlin KR, Lu-Yao G, Malkowicz SB, Mann M, Mille P, Miner MM, Morgan T, Moreno J, Mucci L, Myers RE, Nielsen SM, O'Neil B, Pinover W, Pinto P, Poage W, Raj GV, Rebbeck TR, Ryan C, Sandler H, Schiewer M, Scott EMD, Szymaniak B, Tester W, Trabulsi EJ, Vapiwala N, Yu EY, Zeigler-Johnson C, Gomella LG. Implementation of Germline Testing for Prostate Cancer: Philadelphia Prostate Cancer Consensus Conference 2019. J Clin Oncol. 2020 Aug 20;38(24):2798-2811. doi: 10.1200/JCO.20.00046. Epub 2020 Jun 9. PMID 32516092